CLINICAL TRIAL: NCT04892550
Title: The Addition of a Sagittal Thoracic Posture Corrective Orthotic Device to a Multimodal Rehabilitation Program Improves Management Outcomes in Patients With Chronic Nonspecific Neck Pain: A Randomized-controlled Trial.
Brief Title: Restoring Normal Sagittal Thoracic Posture Improves Management Outcomes in Patients With Chronic Nonspecific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo 2021-5-14
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Rehabilitation
Keywords: Randomized controlled trial; posture; Kyphosis; Neck Pain
MeSH Terms: conditions — Kyphosis; Neck Pain

STUDY DESIGN:
Intervention Model Description: A prospective, parallel-group, randomized clinical trial participants will be randomly assigned to the control group or intervention group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traction group (Experimental): Participants in both groups will complete a 10-week, 3 x per week, 30 sessions total multimodal program consisting of physical pain relief methods, thoracic spine manipulation, myofascial release, and therapeutic exercises.
  In addition, the participants in the intervention group will receive the Denneroll™ thoracic traction orthosis. All participants will begin at 3-minutes per session of DTTO application, each visit they will be encouraged to increase the duration by 2-3 minutes, until such time they will be able to reach the goal of 15-20 minutes per session.
  Interventions: Other: Denneroll traction; Other: Multimodal Program
- Control group (Active Comparator): Participants in both groups will complete a 10-week, 3 x per week, 30 sessions total multimodal program consisting of physical pain relief methods, thoracic spine manipulation, myofascial release, and therapeutic exercises. The multimodal program will be delivered by the same physiotherapist, with 10 years of experience and training in the specific manual techniques in order to minimize inter-therapist variation and enhance fidelity.
  Interventions: Other: Multimodal Program

INTERVENTIONS:
Other: Denneroll traction — The participants will be instructed to lie flat on their back on the ground with their knees slightly bent at 20-30° for comfort and arms gently folded across their stomach. The examiner will position the apex of the Denneroll in one of three regions: lower thoracic (T9-T12), mid-thoracic (T5-T8), and upper-thoracic (T1-T4) depending on the apex of each participant's thoracic kyphosis deformity. For lower thoracic kyphosis (T9-T12) the Denneroll is turned 180° so the peak contacts the lower thoracic spine (T10) while the tapered end supports the mid thoracic region
  Arms: Traction group
Other: Multimodal Program — The multimodal program consists of physical pain relief methods, thoracic spine manipulation, myofascial release, and therapeutic exercises.

SUMMARY:
Because changes in sagittal thoracic alignment have been reported to alter the mechanical loading of the cervical spine and decreased thoracic mobility has been identified as one of the predictors for neck and shoulder pain , it makes sense that thoracic articular treatment improves local kinematics and simultaneously neck pain improves. The purpose of this study is to investigate the effects of a multimodal program, with thoracic hyper kyphosis rehabilitation using the Denneroll™ thoracic traction orthosis , applied to participants with chronic non-specific neck pain and thoracic hyper-kyphosis.

DETAILED DESCRIPTION:
Interventions directed at improving hyper-kyphosis of the thoracic spine may have therapeutic effects on the cervical spine; however, there is a lack of controlled studies evaluating this. The purpose of this study is to investigate the effect effects of a multimodal program, with thoracic hyper kyphosis rehabilitation using the Denneroll™ thoracic traction orthosis , applied to participants with chronic non-specific neck pain and thoracic hyper-kyphosis.

In this study, 80 participants, with chronic non-specific neck pain and thoracic hyper-kyphosis will be included. Participants will be randomly assigned to the control or an intervention group. Both groups will receive the multimodal program; additionally, the intervention group received the Denneroll™ thoracic traction orthosis. Outcome measures will include kyphotic angle (max.), neck pain and disability , sensorimotor control outcomes; head repositioning accuracy , smooth pursuit neck torsion test and overall stability index . Measures will be assessed at three intervals: baseline, 10 weeks, and 6 months after cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* neck pain for more than 3 months
* thoracic angle measured more 55 degrees

Exclusion Criteria:

* Any signs or symptoms of medical "red flags",
* a history of previous spine surgery.
* signs or symptoms of upper motor neuron disease.
* vestibulobasilar insufficiency.
* amyotrophic lateral sclerosis.
* bilateral upper extremity radicular symptoms.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change in thoracic kyphosis | pre-treatment , at 10-week post treatment ,and at 6-month follow up
  Thoracic kyphosis was assessed using a 4D formetric device where determination of thoracic kyphosis angle is measured between tangents from the cervicothoracic junction and that of the thoracolumbar junction

SECONDARY OUTCOMES:
change in neck disability index | pre-treatment , at 10-week post treatment ,and at 6-month follow up
  The neck disability index to assess activities of daily living impact was administered. The NDI has good reliability, validity, and responsiveness to change
Change in numerical rating score | pre-treatment , at 10-week post treatment ,and at 6-month follow up
  Neck pain average intensity over the previous week was assessed using a 0-10 numerical rating score where 0 = no pain, …, 10 = bed ridden and incapacitated.
Change in cervical joint position sense testing | pre-treatment , at 10-week post treatment ,and at 6-month follow up
  Assessment of head repositioning accuracy with the CROM device is performed in an upright seated posture on a stool with no backrest, the CROM device is placed on the participants head, both feet were firmly on the floor with knees bent at an approximate 90° angle. The neutral head position is established as the beginning and reference positions where the CROM device is adjusted to zero for the primary plane of rotational movement. Individuals will be instructed to close their eyes, memorize the starting position, actively rotate their head 30° about the vertical axis, and reposition their head to the starting position with no requirements for speed; only accuracy was encouraged. HRA is measured as the difference in degrees in the primary plane of movement between the origin and the return positions
Change in head and eye movement control: smooth pursuit neck torsion test | pre-treatment , at 10-week post treatment ,and at 6-month follow up
  Electro-oculography will be used for the smooth pursuit neck torsion test to assess disturbances in eye movement control. The test will be performed with the participant's head and trunk in a neutral forward position and then a trunk rotation position (head neutral, trunk in 45° rotation)
Change in Postural Stability | pre-treatment , at 10-week post treatment ,and at 6-month follow up
  Postural stability will be evaluated with a Biodex Balance System . Dynamic balance testing will be assessed allowing simultaneous displacements in both the anterior/posterior and medial/lateral directions

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Diab, professor, Study Director — Cairo Univeristy

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available to other researchers